CLINICAL TRIAL: NCT00006012
Title: Phase I-II Study of Topotecan and Paclitaxel Followed by High-Dose Thoracic Radiation Therapy With Concomitant Cisplatin/Etoposide and Amifostine in Limited-Stage Small Cell Lung Cancer
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Patients With Limited-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N9923; CDR0000068021 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2003-10-08 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Lung Cancer; Radiation Toxicity
Keywords: drug/agent toxicity by tissue/organ; radiation toxicity; limited stage small cell lung cancer
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Lung Neoplasms; Radiation Injuries | interventions — Filgrastim; Amifostine; Cisplatin; Etoposide; Paclitaxel; Topotecan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- topotecan + paclitaxel + filgrastim + TRT + radiation (Experimental): Patients receive topotecan IV on days 1-5 and paclitaxel IV over 3 hours on day 5. Patients receive filgrastim (G-CSF) subcutaneously (SC) daily beginning 24 hours after the last dose of chemotherapy and continuing until blood counts recover. Treatment repeats every 3 weeks for 2 courses.
  After 2 courses of treatment, patients undergo TRT twice daily for 5 consecutive days for 5 weeks. During TRT, patients receive cisplatin IV, oral etoposide, and amifostine SC daily prior to TRT.
  At 4 weeks after completion of TRT, patients receive 2 additional courses of topotecan, paclitaxel, and G-CSF every 3 weeks followed by prophylactic cranial irradiation.
  Patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 3 years.
  Interventions: Biological: filgrastim; Drug: amifostine trihydrate; Drug: cisplatin; Drug: etoposide; Drug: paclitaxel; Drug: topotecan hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
Drug: amifostine trihydrate
Drug: cisplatin
Drug: etoposide
Drug: paclitaxel
Drug: topotecan hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy before, during, and after radiation therapy in treating patients who have limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of thoracic radiotherapy administered with cisplatin, etoposide, and amifostine preceded and followed by topotecan and paclitaxel in patients with limited stage small cell lung cancer (phase I closed to accrual as of 5/27/2004).
* Determine the two-year survival of this patient population treated with this regimen.
* Determine the two-year, progression-free local control rate in this patient population treated with this regimen.
* Assess the tolerability of this treatment regimen in these patients.
* Determine the antitumor activity of this regimen in these patients.
* Determine the overall survival and overall time to progression in this patient population treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of thoracic radiotherapy (TRT).

Patients receive topotecan IV on days 1-5 and paclitaxel IV over 3 hours on day 5. Patients receive filgrastim (G-CSF) subcutaneously (SC) daily beginning 24 hours after the last dose of chemotherapy and continuing until blood counts recover. Treatment repeats every 3 weeks for 2 courses.

After 2 courses of topotecan and paclitaxel, patients undergo TRT twice daily for 5 consecutive days for 5 weeks. During TRT, patients receive cisplatin IV, oral etoposide, and amifostine SC daily prior to TRT.

At 4 weeks after completion of TRT, patients receive 2 additional courses of topotecan, paclitaxel, and G-CSF every 3 weeks followed by prophylactic cranial irradiation.

Cohorts of 3-6 patients receive escalating doses of TRT until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity (phase I closed to accrual as of 5/27/2004).

Patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 3-73 patients will be accrued for this study (phase I closed to accrual as of 5/27/2004).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer
* Limited disease confined to one hemithorax, the ipsilateral supraclavicular fossa, and encompassable within tolerable thoracic radiotherapy field

  * Minimal pleural effusions (i.e., blunting of the costophrenic angle on chest x-ray or a small effusion on CT scan) allowed
* Measurable disease

  * At least one lesion accurately measured in at least 1 dimension with longest diameter at least 20 mm

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 3 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Pulmonary:

* FEV_1 at least 40% of predicted AND at least 1 liter

Other:

* No uncontrolled infection
* No other severe underlying diseases
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or noninvasive carcinomas (carcinoma in situ)
* No grade 2 or greater peripheral neuropathy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No hypersensitivity to E.coli-derived proteins, filgrastim (G-CSF), or any excipients of G-CSF

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No prior hemithorax radiotherapy

Surgery

* Not specified

Other

* No prior therapy for small cell lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2001-02; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Survival at 2 years | at 2 years

SECONDARY OUTCOMES:
Local progression-free survival at 2 years | at 2 years
Overall survival | Up to 5 years
Time to progression | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Okuno, MD, Study Chair — Mayo Clinic
Locations (84):
- United States (84):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Bryan LGH Medical Center West, Lincoln, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - St. Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P.C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Franciscan Skemp Healthcare, La Crosse, Wisconsin

REFERENCES:
- [Result] Garces YI, Okuno SH, Schild SE, Mandrekar SJ, Bot BM, Martens JM, Wender DB, Soori GS, Moore DF Jr, Kozelsky TF, Jett JR. Phase I North Central Cancer Treatment Group Trial-N9923 of escalating doses of twice-daily thoracic radiation therapy with amifostine and with alternating chemotherapy in limited stage small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2007 Mar 15;67(4):995-1001. doi: 10.1016/j.ijrobp.2006.10.034. PMID 17336213
- [Result] Garces YI, Okuno SH, Schild SE, et al.: A phase I/II NCCTG trial of escalating doses of twice daily thoracic radiation therapy (TRT) in limited-stage small cell lung cancer (LSCLC). [Abstract] J Clin Oncol 23 (Suppl 16): A-7163, 661s, 2005.